CLINICAL TRIAL: NCT06951906
Title: Imaging Biomarkers of Freezing of Gait Response to Deep Brain Stimulation
Brief Title: Imaging Biomarkers of FOG Response to DBS
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Gonzalo Revuelta, Associate Professor of Neurology, Medical University of South Carolina
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00131410; 1R01NS131396-01A1 (NIH)
Record Dates: First submitted 2025-04-23; First posted 2025-04-30 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Freezing of Gait Symptoms in Parkinson's Disease; Deep Brain Stimulation
Keywords: Freezing of Gait; Parkinson's Disease; Deep Brain Stimulation
MeSH Terms: conditions — Parkinson Disease | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- PD Patients with FOG undergoing DBS (Active Comparator)
  Interventions: Diagnostic Test: fMRI

INTERVENTIONS:
Diagnostic Test: fMRI — Baseline imaging will utilize advanced diffusion MRI metrics to determine which brain areas are structurally connected to the stimulation target and their structural integrity. Post-operative assessments will include behavioral measures of FOG response and imaging measures of neural response to stimulation. Pre- and post-operative data will be used to evaluate the association between structural integrity, connectivity and behavioral response.

SUMMARY:
For this study, the investigators are recruiting 54 individuals with Parkinson's Disease and Freezing of Gait (FOG) who are planning to undergo Deep Brain Stimulation (DBS). The objective of this study is to better understand the FOG response to DBS. Prior to DBS, participants will undergo an MRI scan, behavioral assessment related to walking, a cognitive evaluation, and assessment of other Parkinson's disease symptoms. Following DBS, participants will repeat these assessments at multiple timepoints over the period of one year. Overall, participants will complete a total of 7 visits over a period of approximately 1 year.

DETAILED DESCRIPTION:
The long-term goal of this research is to develop an individualized approach for the treatment of Freezing of Gait (FOG) with Deep Brain Stimulation (DBS). In pursuit of this goal, the investigators have preliminary findings which show that:

1. Effective subthalamic nucleus DBS (STN-DBS) activates the globus pallidus interna (GPi) and decreases cortical activation in Parkinson's Disease (PD);
2. Structural connectivity to the GPi, supplemental motor area (SMA), and primary motor cortex (M1) is associated with DBS response in FOG; and
3. Decreased microstructural integrity of the GPi is associated with decreased DOPA response in FOG.

The investigators propose a conceptual framework whereby engaging a specific FOG response network depends on the structural integrity of the network, as well as lead placement and stimulation parameters. The investigators propose to recruit 54 individuals with FOG who are identified as appropriate STN-DBS candidates to undergo a prospective longitudinal imaging and behavioral study of FOG response to STN-DBS. Baseline behavioral assessments will characterize FOG behavior, severity, subtype, as well as the cognitive profile, non-FOG motor severity, and other demographics of the enrolled participants that may contribute to DBS response. Baseline imaging will utilize advanced diffusion MRI metrics to determine which brain areas are structurally connected to the stimulation target and their structural integrity. Post-operative assessments will include behavioral measures of FOG response and imaging measures of neural response to stimulation. Pre- and post-operative data will be used to evaluate the association between structural integrity, connectivity, and behavioral response.

ELIGIBILITY:
Inclusion Criteria:

1. >40 years of age.
2. diagnosis of PD based on UK Brain Bank diagnostic criteria.
3. presence of FOG, defined as a score of 1 on part 1 of the nFOGQ and confirmed by objective evaluation (a score of 1 represents a positive response of having experienced such an episode over the last month).
4. clinically selected at the MUSC DBS Conference to undergo STN-DBS surgery.

Exclusion Criteria:

1. a history of other significant gait impairment unrelated to PD (e.g. orthopedic deformities).
2. inability to complete gait assessments (timed-up-and-go task) in the OFF state without assistance or assist devices.
3. contraindications to MRI, including inability to lie supine in the scanner environment, pregnancy, and non-MRI compatible metal implants.
4. implantation of non-3 T MRI-compatible DBS devices.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-11-11 (Actual); Primary Completion 2029-11 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Turn Duration | Assessed at Baseline (Visit 3) and at 12 months post-activation (Visit 7)
  Turn duration is measured during the timed up and go (TUG) task. Subjects are instrumented with inertial measurement units (IMUs), and turn duration is measured from the first step onto a marked box to the last toe off the box during the turn.
Difference in BOLD Response to STN-DBS | Assessed post-operatively at 6 months (Visit 5) and 12 months (Visit 6).
  Whole-brain activation is assessed via BOLD signal changes associated with T2*-relaxation rate during combined Deep Brain Stimulation and functional MRI (DBS-fMRI). This involves cycling the DBS device ON and OFF during resting-state scans
Difference in Structural Connectivity | Based on baseline diffusion MRI data (Visit 4) and analyzed in relation to DBS response determined at 12 months post-activation.
  Structural connectivity profiles are determined using individual structural connectivity data and the Volume of Tissue Activated (VTA) model, which accounts for stimulation settings and lead placement. The outcome is the comparison of VTA connectivity to specific brain regions (e.g., GPi, SMA, M1, GPe) between STN-DBS responsive and unresponsive participants.
Difference in Structural Integrity | Based on baseline diffusion MRI data (Visit 4) and analyzed in relation to DBS response determined at 12 months post-activation.
  Microstructural integrity of brain structures (e.g., STN, GPi, PPN) is assessed using advanced diffusion MRI metrics, specifically Diffusional Kurtosis Imaging (DKI). The outcome is the comparison of these metrics between STN-DBS responsive and unresponsive participants.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1. Forsaa EB, Larsen JP, Wentzel-Larsen T, Alves G. A 12-year population-based study of freezing of gait in Parkinson's disease. Parkinsonism Relat Disord 2015; 21(3): 254-8. 2. Perez-Lloret S, Negre-Pages L, Damier P, et al. Prevalence, determinants, and effect on quality of life of freezing of gait in Parkinson disease. JAMA Neurol 2014; 71(7): 884-90. 3. Nieuwboer A, Giladi N. Characterizing freezing of gait in Parkinson's disease: Models of an episodic phenomenon. Mov Disord 2013; 28(11): 1509-19. 4. Nutt JG, Bloem BR, Giladi N, Hallett M, Horak FB, Nieuwboer A. Freezing of gait: moving forward on a mysterious clinical phenomenon. Lancet Neurol 2011; 10(8): 734-44. 5. Moore O, Peretz C, Giladi N. Freezing of gait affects quality of life of peoples with Parkinson's disease beyond its relationships with mobility and gait. Mov Disord 2007; 22(15): 2192-5. 6. Grimbergen YA, Munneke M, Bloem BR. Falls in Parkinson's disease. Curr Opin Neurol 2004; 17(4): 405-15. 7. Walton CC, Shine JM, Hall JM, et al. The major impact of freezing of gait on quality of life in Parkinson's disease. J Neurol 2015; 262(1): 108-15. 8. Barbe MT, Tonder L, Krack P, et al. Deep Brain Stimulation for Freezing of Gait in Parkinson's Disease With Early Motor Complications. Mov Disord 2020; 35(1): 82-90. 9. Defer GL, Widner H, Marie RM, Remy P, Levivier M. Core assessment program for surgical interventional therapies in Parkinson's disease (CAPSIT-PD). Mov Disord 1999; 14(4): 572-84. 10. Artusi CA, Lopiano L, Morgante F. Deep Brain Stimulation Selection Criteria for Parkinson's Disease: Time to Go beyond CAPSIT-PD. J Clin Med 2020; 9(12). 11. Charles PD, Van Blercom N, Krack P, et al. Predictors of effective bilateral subthalamic nucleus stimulation for PD. Neurology 2002; 59(6): 932-4. 12. Welter ML, Houeto JL, Tezenas du Montcel S, et al. Clinical predictive factors of subthalamic stimulation in Parkinson's disease. Brain 2002; 125(Pt 3): 575-83. 13. Schlenstedt C, Shalash A, Muthuraman M, Fal
- See also: Investigating Gait with NeuroImaging & Neuromodulation — https://medicine.musc.edu/departments/neurology/research/ignition-lab